CLINICAL TRIAL: NCT03751800
Title: An Observational, Prospective, Multicentre Study to Assess the Sensitivity to Change of the SAMANTA Questionnaire in Women with Heavy Menstrual Bleeding (HMB)
Brief Title: A Study Run At Multiple Study Sites to Test Whether the SAMANTA Questionnaire That is Used to Diagnose Heavy Menstrual Bleeding (HMB), Can Also Be Used to Assess Changes of Severity of HMB in Women with HMB Who Are Treated During 12 Months with a Chronic Hormonal Treatment
Acronym: SAMIRA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20061
Record Dates: First submitted 2018-11-21; First posted 2018-11-23 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Menorrhagia
Keywords: Heavy Menstrual Bleeding
MeSH Terms: conditions — Menorrhagia | interventions — Estradiol; dienogest; Medroxyprogesterone Acetate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with HMB: Women with a diagnostic of HMB according to medical criteria and based on clinical judgment that have freely chosen a chronic hormonal treatment under therapeutic indication of HMB in Spain
  Interventions: Drug: Chronic hormonal treatment

INTERVENTIONS:
Drug: Chronic hormonal treatment — Drugs used in this study are described by the physicians during routine gynecological visits
  Other Names: 1. Mirena (Levonorgestrel - IUS); 2. Qlaira (Estradiol valerate and dienogest); 3. Progevera (Medroxyprogesterone acetate); and any new hormonal treatment marketed in Spain that has the indication for HMB

SUMMARY:
A study run at multiple study sites in Spain to test whether the SAMANTA questionnaire that is used to diagnose heavy menstrual bleeding (HMB), can also be used to assess changes of severity of HMB in women with HMB who are treated during 12 months with a chronic hormonal treatment. Patients that are treated with chronic hormonal treatment as Levonorgestrel (trade name Mirena) or with a combination of estradiol valerate and dienogest (trade name Qlaira) or with Medroxyprogesterone acetate (trade name Progevera) and any new hormonal treatment marketed in Spain that has the indication for HMB in routine gynaecological practice are observed for 12 months in this study or for a shorter period in time in case of withdrawal. The study aims also to describe the overall satisfaction of women with their chronic hormonal treatment for HMB and how the women think their menstrual bleeding has changed. In addition the study aims to describe the changes of the score that is derived from the SAMANTA questionnaire in relation to Quality of Life. Quality of Life is measured with the SF36v2 questionnaire. The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health.

ELIGIBILITY:
Inclusion Criteria:

* Women in childbearing age, ≥18 years old, not intending to become pregnant during the next year.
* Women diagnosed with heavy menstrual bleeding or idiopathic menorrhagia according to medical criteria and based on clinical judgment.
* Women for whom the clinician decides, in agreement with the patient, to prescribe any of the available chronic hormonal treatments with the therapeutic indication of HMB in Spain (Mirena, Qlaira or Progevera).
* Women capable of reading and writing.
* Women who signed the informed consent.

Exclusion Criteria:

* Women with amenorrhea or menopause.
* Women with contraindications and warnings with the chronic hormonal treatment prescribed for HMB as per the summary of product characteristics (interaction with concomitant medication, etc.).
* Women receiving contraceptive hormonal therapy or using a copper intrauterine device.
* Women on hormone replacement therapy.
* Women with a history of malignancy.
* Women with degenerative diseases that could directly negatively impact their daily life.
* Women who have given birth within the previous 6 months.
* Women who are pregnant.
* Women participating in an investigational program with interventions outside of routine clinical practice.
* Women with psychiatric disorders who are unable to make decisions and follow instructions.
* Women with concomitant medication that may lead to changes in the bleeding pattern (e.g. antiplatelet and/ or anticoagulants).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women in childbearing age, with diagnosed HMB according to medical criteria and based on clinical judgment and for whom the clinician decides, in agreement with the patient, to prescribe a chronic hormonal treatment with the therapeutic indication of HMB or idiopathic menorrhagia (IM) in Spain during a routine gynaecological visit.
Sampling Method: Probability Sample
Enrollment: 422 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
SAMANTA questionnaire score | Up to 12 months
  SAMANTA questionnaire: is a existing and validated tool has shown that it can be effectively used by gynaecologists to easily discriminate among women with and without HMB

SECONDARY OUTCOMES:
Overall satisfaction with the chronic hormonal treatment measured with a user satisfaction questionnaire | Up to 12 months
Changes in menstrual bleeding pattern measured with a user satisfaction questionnaire | Up to 12 months
Correlation between changes in SAMANTA score and changes in women's quality of life measured with SF36v2 questionnaire | Up to 12 months
  SF36v2: Generic health questionnaire, which comprises five dimensions: mobility, self-care, usual activities, pain/ discomfort and anxiety/ depression

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Many Locations, Spain

REFERENCES:
- [Background] Perello-Capo J, Rius-Tarruella J, Andeyro-Garcia M, Calaf-Alsina J. Sensitivity to Change of the SAMANTA Questionnaire, a Heavy Menstrual Bleeding Diagnostic Tool, After 1 Year of Hormonal Treatment. J Womens Health (Larchmt). 2023 Feb;32(2):208-215. doi: 10.1089/jwh.2022.0155. Epub 2022 Dec 22. PMID 36576860
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/